CLINICAL TRIAL: NCT05715606
Title: Safety and Efficacy of Metabolically Armed CD19 CAR-T Cells (Meta10-19) in the Treatment of r/r DLBCL Clinical Research
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Leman Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Meta10-19-001
Record Dates: First submitted 2022-12-27; First posted 2023-02-08 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Meta10-19; CAR-T Cells Therapy; r/r DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of Metabolically Armed CD19 CAR-T cells (Experimental): Patients undergo leukapheresis. Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CAR-T cells infusion. A dose of metabolically armed CD19 CAR-T cells will be infused on day 0.
  Interventions: Drug: Metabolically Armed CD19 CAR-T cells

INTERVENTIONS:
Drug: Metabolically Armed CD19 CAR-T cells — Each subject receive metabolically armed CD19 CAR-T cells by intravenous infusion
  Other Names: Meta10-19

SUMMARY:
A Study of Metabolically Armed CD19 CAR-T Cells Therapy for Patients With Relapsed and/or Refractory Diffuse Large B-Cell Lymphoma

DETAILED DESCRIPTION:
This is a single arm, open-label study. This study is indicated for relapsed or refractory CD19+ Diffuse Large B-Cell Lymphoma. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products.

1. Main research objectives:

   To evaluate the safety and efficacy of metabolically armed CD19 CAR-T Cells in the treatment of r/r DLBCL.
2. Secondary research objectives:

（1）To evaluate the pharmacokinetic (PK) and pharmacodynamics(PD) characteristics of metabolically armed CD19 CAR-T Cells after infusion.

（2）To evaluate tumor remission after infusion of metabolically armed CD19 CAR-T Cells.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her guardian voluntarily signed the informed consent;
2. Adult Patients with relapsed and refractory diffuse large B-cell lymphoma (Primary mediastinal large B-cell lymphoma and transformed follicular lymphoma are included)

   Definition of refractory:
   1. No response to the last treatment, including:

      The best response to the last treatment was PD, or ; The best response to the last treatment was SD and the duration was not more than 6 months after the last dose.
   2. Not suitable for autologous hematopoietic stem cell transplantation (ASCT), or ASCT refractory, including:

   Disease progression or recurrence within 12 months or less (recurrence must be confirmed by biopsy) after ASCT treatment, or; Patients accept remedial treatment after ASCT must have no response or relapse after the last treatment.
3. Patients who had previously received ≥2 lines therapy including at least:

   1. A chemotherapy regimen containing anthracyclines；
   2. For patients with transformed DLBCL from follicular lymphoma, they must have previously received chemotherapy for follicular lymphoma and have refractory disease after transformation to DLBCL.
4. CD19 expression was positive by immunohistochemistry or flow cytometry (accept the results of this peripheral blood mononuclear cells or previous report from a Class A tertiary hospital before peripheral blood collection)
5. At least one measurable lesion at baseline, according to the initial assessment, staging and Response Assessment recommendations for Hodgkin's and non-Hodgkin's lymphoma (2014 edition)
6. Expected survival time greater than 12 weeks
7. The baseline ECOG score was 0 or 1
8. organ function：

   1. Kidney function is defined as:

      Serum creatinine ≤1.5 times ULN, or； The glomerular filtration rate (eGFR) estimated by MDRD formula was ≥60m/min/1.73m2；[eGFR=186×（age）-0.203×SCr-1.154（mg/dl），for females, the result was ×0.742]；
   2. Liver function is defined as： ALT≤5 times ULN, and; Patients with total bilirubin ≤2.0mg/dl, except those with Gilbert-Meulengracht syndrome. Patients with Gilbert-.Meulengracht syndrome with total bilirubin ≤3.0 times ULN and direct bilirubin ≤1.5 times ULN were included.
   3. Pulmonary function: ≤CTCAE grade 1 dyspnea and oxygen saturation of blood (SaO2) ≥91% in indoor air environment.
9. Hemodynamic stability was determined by echocardiography or multichannel radionuclide angiography (MUGA) and LVEF ≥45％
10. Patients using the following drugs must meet the following conditions:

    1. Steroid: Therapeutic doses of steroids must be discontinued 2 weeks prior to Meta10-19 infusion. However, physiological replacement doses of steroids are permitted, hydrocortisone or its equivalent < 6-12mg/mm2/ day；
    2. Immunosuppressive agent: Any immunosuppressive drug must be stopped ≥4 weeks before the informed consent is signed
    3. Anti-proliferative therapy in addition to preconditioning chemotherapy 2 weeks prior to Meta10-19 infusion
    4. Treatment for CNS disease must be stopped 1 week before Meta10-19 infusion (e.g., intrathecal methotrexate)
11. The patient has recovered from the toxicity of the previous treatment, that is, the CTCAE toxicity grade is less than 1 (The exception is specific toxicity of grade 2 or less, such as hair loss, which the researchers have determined is not recoverable in a short period of time) is suitable for pretreatment chemotherapy and CAR T cell therapy
12. Women of childbearing age and all male patients must consent to use a effective contraception for at least 12 months after Meta10-19 infusion and until two consecutive PCR tests show no more CAR T cells in vivo；

Exclusion Criteria:

1. Patients with present or history of central nervous system diseases such as seizures disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
2. Patients with history of allogeneic hematopoietic stem cell transplantation
3. Patients who had received chemotherapy other than preconditioning chemotherapy within 2 weeks prior to Meta10-19 infusion
4. Patients who participated in other clinical trials within 30 days prior to enrollment
5. Patients with active hepatitis B (defined as hepatitis B surface antigen positive or hepatitis B core antibody positive, concomitant hepatitis B virus DNA level > 1000 copies/ml) or hepatitis C (HCV RNA positive)
6. Patients with HIV antibody positive or treponema pallidum antibody positive
7. Patients with uncontrolled acute life-threatening bacterial, viral or fungal infections (e.g. positive blood cultures ≤72 hours before Meta10-19 infusion)
8. Patients with unstable angina pectoris and/or myocardial infarction within 6 months prior to enrollment
9. Patients with history of other malignancies, but the following conditions can be enrollment:

   1. Adequately treated basal or squamous cell carcinoma (requiring adequate wound healing before signing informed consent);
   2. Carcinoma in situ (DCIS) of cervical or breast cancer, which has been treated therapeutically, has shown no signs of recurrence for at least 3 years prior to the signing of the informed consent；
   3. The primary malignancy has been completely resected and in complete remission for ≥5 years；
10. Women who are pregnant or breastfeeding (pregnancy tests for women of childbearing age are positive)
11. Patients with active neuroautoimmune or inflammatory conditions (e.g. Guillian-Barre syndrome, amyotrophic lateral sclerosis);
12. Other conditions that the investigator considered should not be enrolled in this clinical study, such as poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
MTD | MTD will be determined based on DLTs observed during the first 28 days of study treatment.
  Determine the Maximal Tolerable Dose(MTD)
Objective response rate (ORR) | Within 3 months following infusion of Meta10-19
  Measure Tumor response rate (including CR and PR) .

SECONDARY OUTCOMES:
Pharmacokinetics | Up to 12 months after CAR-T treatment
  The number of CAR-T cells in peripheral blood was measured to evaluate the persistence of CAR-T cells
Pharmacodynamics | Up to 28 days after infusion
  Peak level of cytokines in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No